CLINICAL TRIAL: NCT02518802
Title: Pemetrexed Disodium and Cisplatin Chemotherapy Combined With Synchronous Gefitinib vs Chemotherapy Alone as Adjuvent Therapy in Patient With Stage II-IIIA, Epidermal Growth Factor Receptor Mutant Expressing Lung Adenocarcinoma
Brief Title: Pemetrexed Combined With Synchronous Gefitinib as Adjuvent Therapy in Patient With EGFR Mutant Lung Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W-TONG002
Record Dates: First submitted 2015-05-05; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-04

CONDITIONS: Lung Neoplasms
Keywords: Gefitinib; Pemetrexed; Synchronous therapy; Adjuvent therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Gefitinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synchronous therapy (Experimental): 'Gefitinib and Pemetrexed' Synchronous use of Gefitinib for 2 years during or after chemotherapy with Pemetrexed plus Cisplatin regimen. Gefitinb, 250mg per day,take orally for 2 years. Pemetrexed, 500mg/m2, day 1; Cisplatin 75mg/m2, day 1. Three weeks as a cycle. Four cycles in total.
  Interventions: Drug: Gefitinib; Drug: Pemetrexed
- Chemotherapy (Active Comparator): Pemetrexed: Pemetrexed, 500mg/m2, day 1; Cisplatin 75mg/m2, day 1. Three weeks as a cycle. Four cycles in total.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250mg per day for 2 years.
  Other Names: Iressa
  Arms: Synchronous therapy
Drug: Pemetrexed — Pemetrexed, 500mg/m2, day 1; Cisplatin 75mg/m2, day 1. Three weeks as a cycle. Four cycles in total.
  Other Names: Alimta

SUMMARY:
This randomized phase III trial is studying gefitinib and synchronous pemetrexed/cisplatin chenmotherapy to see how well it works compared to pemetrexed/cisplatin chenmotherapy alone in treating patients who have undergone surgery for stage II-IIIA(N1-N2) lung adenocarcinoma with EGFR activating mutation in Asian population.

DETAILED DESCRIPTION:
Adjuvant cisplatin-based chemotherapy is recommended for routine use in patients with stages IIA, IIB, and IIIA non-small cell lung cancer (NSCLC) after complete resection. Cisplatin and pemetrexed combination is the standard regimen for lung adenocarcinoma in adjuvant setting. The BR. 19 trial reported adjuvant gefitinib after complete resection of early stage NSCLC(stage IB 49%, II 38%, III 13%) did not confer disease free survival(DFS) or overall survival(OS) advantage in overall population. While the median gefitinib treatment time is only 4.8 months. There are only 76 patients with EGFR mutations included in this analysis. The study closed prematurely in 2005.

Activating somatic mutations of the tyrosine kinase domain of epidermal growth factor receptor (EGFR) have been characterized in a subset of patients with advanced NSCLC.The EGFR mutation rate was 30% in Chinese NSCLC. Patients harboring these mutations in their tumors show excellent response to EGFR tyrosine kinase inhibitors (EGFR-TKIs). This randomized phase III trial is studying gefitinib and synchronous pemetrexed/cisplatin chenmotherapy to see how well it works compared to pemetrexed/cisplatin chenmotherapy alone in treating patients who have undergone surgery for stage II-IIIA(N1-N2) lung adenocarcinoma with EGFR activating mutation in Asian population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males or females aged ≥18 years, < 70 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Target population is completely resected pathological stage II-IIIA(N1-N2) NSCLC with EGFR exon 19 deletions and exon 21 L858R activating mutation.
* Patient who can start the investigational therapy within 3-6 weeks after the complete resection
* ECOG performance status 0-1.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Known severe hypersensitivity to gefitinib or any of the excipients of this product.
* Known severe hypersensitivity to pre-medications required for treatment with cisplatin / vinorelbine doublet chemotherapy.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* Interstitial pneumonia.
* Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy).
* Patients with prior radiotherapy
* History of another malignancy in the last 5 years with the exception of the following:Other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Eye inflammation or eye infection not fully treated or conditions predisposing the subject to this.
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.
* Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over)
* Patients who harbouring exon 20 T790M mutation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From date of randomization to the first documented disease progression or death, whichever occurs first, assessed up to 3 and 5 years.
  To evaluate the disease free survival of synchronous therapy versus combination of Pemetrexed plus Cisplatin as adjuvant treatment for pathological stage II-IIIA(N1-N2) lung adenocarcinoma with EGFR mutation.Disease free survival (DFS)- defined as the time from randomization to the first documented disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | From date of randomization to the first documented death, assessed up to 5 years.
  To evaluate the overall survival of synchronous therapy versus combination of Pemetrexed plus Cisplatin as adjuvant treatment for stage II-IIIA(N1-N2) lung adenocarcinoma with EGFR mutation.
Number of Participants with Adverse Events | In the period of Gefitinib 250 mg/day oral daily for 24 months. Pemetrexed 500 mg/m2 intravenous infusion on day 1, Cisplatin 75 mg/m2 on day 1 for 4 cycles.
  The safety and tolerability profile of gefitinib at a 250 mg daily dose relative to that of Chemotherapy.
Quality of life | In the period of Gefitinib 250 mg/day oral daily for 24 months. Pemetrexed 500 mg/m2 intravenous infusion on day 1, Cisplatin 75 mg/m2 on day 1 for 4 cycles.
  Quality of life as measured by the total score and Trial Outcome Index (TOI) of the Functional Assessment of Cancer Therapy - Lung Cancer (FACT-L) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Li Xiaofei, MD, Principal Investigator — Tangdu Hospital of the Fourth Millitary Medical University; Yan Xiaolong, MD, Study Director — Tangdu Hospital of the Fourth Millitary Medical University
Locations (1):
- Tangdu Hospital of the Fourth Millitary Medical University, Xi'an, Shaanxi, China